CLINICAL TRIAL: NCT06764732
Title: Laser Assisted Socket Seal Surgery Using Bioactive Glass for Dental Implant Site Development
Brief Title: Socket Seal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nora Abdelgawad Mohamed, associate professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DU:024100558
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2022-11

CONDITIONS: Socket Sealing
Keywords: bio active glass; socket preservation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): platelet rich fibrin membrane
  Interventions: Biological: Platelet rich fibrin
- test 1 group (Experimental): bioactive glass
  Interventions: Biological: bioactive glass; Biological: Platelet rich fibrin
- test 2group (Active Comparator): bioactive glass and Photobiomodulation
  Interventions: Biological: bioactive glass; Radiation: bioactive glass graft and PBM irradiation; Biological: Platelet rich fibrin

INTERVENTIONS:
Biological: bioactive glass — supplied as resorbable form, (400-800um) particle siz
  Arms: test 1 group; test 2group
Radiation: bioactive glass graft and PBM irradiation — The used laser parameters were set as: wavelength, 980 nm; power, 0.55 W; energy, 36 J; power density, 0.76 W cm2
  Arms: test 2group
Biological: Platelet rich fibrin — 10 ml of blood was withdrawn from the patient and immediately centrifuged for 10 minutes at 3000 revolutions/min and the layer of fibrin clot was obtained

SUMMARY:
laser photo biomodulation (PBM) as a supplement to socket seal surgery

DETAILED DESCRIPTION:
the role of PBM therapy as an adjunct for bioactive glass graft in SSS approaches

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least a periodontal-affected and non-restorable tooth in posterior region (Class II sockets).
* At least 10% plaque control scoring was accepted
* A moderate to thick gingival phenotype

Exclusion Criteria:

* systemic diseases or conditions that may compromise healing or bone metabolism,
* having a history of radiotherapy, chemotherapy or bisphosphonate therapy, previous use of antibiotics in the last 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
alveolar ridge dimensional changes in height and width measures | at base line and after 9 months

SECONDARY OUTCOMES:
bone biopsy | after 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- , Faculty of Oral and Dental Medicine, Delta University for Science and Technology (DU), Dakahlia, Egypt, Dakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hazzaa HH, Shiekh MAME, AbdAllah MF, Abdelgawad N, El-Mahdy MA, Shoshan HS, Elewa GM. Laser-assisted socket seal surgery using bioactive glass for dental implant site development: a randomized clinical trial. Sci Rep. 2025 Dec 9;15(1):43386. doi: 10.1038/s41598-025-28824-7. PMID 41360883
- See also: Related Info — https://doi.org/10.5051/jpis.2005120256